CLINICAL TRIAL: NCT04106661
Title: Tai Chi Via DVD Instruction as an Introduction to Physical Activity for Women With Morbid Obesity: a Feasibility Study
Brief Title: Tai Chi as Physical Activity for Women With Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Husson University (Other)
Responsible Party: Principal Investigator, Cathy Stucker, Assistant Professor, Husson University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16PT03; 16-1-M-325 (Other: Eastern Maine Medical Center)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Morbid Obesity
Keywords: Tai Chi; physical activity; morbid obesity
MeSH Terms: conditions — Obesity, Morbid; Motor Activity | interventions — Tai Ji; Exercise

STUDY DESIGN:
Intervention Model Description: Pretest-posttest control group design: The groups were determined by convenience sample due to the time-sensitive need to form the exercise groups. There were two arms of the study that aligned with two concurrent academic years. The first six participants to express interest were placed in the first Tai Chi intervention group. The next three participants were in the first control group. The second arm of the study had five participants who made contact before the second exercise group began. The second control group had three participants.
Who Masked: Outcomes Assessor
Masking Description: Data was de-identified prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Intervention 1 (Experimental): The intervention group and control group were recruited during the same time frame. The intervention group received Tai Chi instruction via a weekly group session and home use of a DVD. The control group received no formal instruction in physical activity.
  Interventions: Other: Tai Chi
- Tai Chi Intervention 2 (Experimental): The intervention group and control group were recruited during the same time frame. The intervention group received Tai Chi instruction via a weekly group session and home use of a DVD. The control group received no formal instruction in physical activity.
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Tai Chi — Physical activity requiring slow, controlled whole body movement and weight shifting.
  Other Names: physical activity

SUMMARY:
This study investigated the use of Tai Chi as a feasible form of physical activity for women with morbid obesity utilizing an instructional digital video disc (DVD). Two groups of women with morbid obesity (body mass index of >40) were placed into the Tai Chi intervention group or the control group. Initial function was assessed with a series of tests and then repeated after 8 weeks. During the 8 weeks, the Tai Chi intervention group met once a week for 45 minutes to participate in a group exercise class. The control group was asked to continue their regular activity. At the end of the 8 weeks, both groups were reassessed with the same tests from the start of the study. The investigators hypothesized that the Tai Chi group would show more improvement in their functional scores for strength, balance and quality of life than the control group.

DETAILED DESCRIPTION:
The purpose of this study was to investigate an alternative approach to physical activity in people who are morbidly obese to improve their overall health, functional mobility, and quality of life. Although physical activity is recommended in most weight management programs, the type of physical activity that results in the most successful outcomes has not been determined. Walking programs are among the most common forms recommended, however few parameters or guidelines are provided, and well-controlled comparisons to other types of exercise are lacking. Compliance with exercise programs is also a factor that impacts success, therefore offering solutions that improve compliance would be beneficial as well. This study investigated the use of home-based exercise enhanced with DVDs along with weekly, supervised group sessions to compare Tai Chi to a walking program in participants who are morbidly obese.

The participants were recruited from the community with the requirement that they have a body mass index of >40 and have a diagnosis of morbid obesity. A falls risk screening, the Four Square Step Test (FSST), was performed on which they must score as a low fall risk. A battery of physical and paper tests will be completed prior to starting the study to assess balance, endurance, functional lower extremity strength, and quality of life. Both groups completed a self-report of their weekly physical activity that was submitted on an Activity Log. Those who were designated to be in the control group did not have any additional interaction with the study until week 10 when they returned for post-testing. The Tai Chi intervention group met one time per week as a group to practice Tai Chi with the DVD as the guide. Physical therapy students and faculty were present at each session to modify and supervise as needed. The intervention group also followed the DVD in the home setting for 2 additional sessions each week. Following the 8 weeks of structured classes and home activity, the participants returned the following week for the post-testing session.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than 40
* Completion of the four square step test in less than 15 seconds.

Exclusion Criteria:

* History of neurological insult or disease
* Cardiac condition limiting exercise
* Joint pain severely limiting movement
* Major surgery within 6 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Stucker, DSc, Principal Investigator — Husson University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Kahn EB, Ramsey LT, Brownson RC, Heath GW, Howze EH, Powell KE, Stone EJ, Rajab MW, Corso P. The effectiveness of interventions to increase physical activity. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):73-107. doi: 10.1016/s0749-3797(02)00434-8. PMID 11985936
- [Background] Puhl R, Suh Y. Health Consequences of Weight Stigma: Implications for Obesity Prevention and Treatment. Curr Obes Rep. 2015 Jun;4(2):182-90. doi: 10.1007/s13679-015-0153-z. PMID 26627213
- [Background] Liu X, Vitetta L, Kostner K, Crompton D, Williams G, Brown WJ, Lopez A, Xue CC, Oei TP, Byrne G, Martin JH, Whiteford H. The effects of tai chi in centrally obese adults with depression symptoms. Evid Based Complement Alternat Med. 2015;2015:879712. doi: 10.1155/2015/879712. Epub 2015 Jan 21. PMID 25688280
- [Background] Lachman S, Boekholdt SM, Luben RN, Sharp SJ, Brage S, Khaw KT, Peters RJ, Wareham NJ. Impact of physical activity on the risk of cardiovascular disease in middle-aged and older adults: EPIC Norfolk prospective population study. Eur J Prev Cardiol. 2018 Jan;25(2):200-208. doi: 10.1177/2047487317737628. Epub 2017 Nov 21. PMID 29161890
- [Background] Jagielski AC, Brown A, Hosseini-Araghi M, Thomas GN, Taheri S. The association between adiposity, mental well-being, and quality of life in extreme obesity. PLoS One. 2014 Mar 26;9(3):e92859. doi: 10.1371/journal.pone.0092859. eCollection 2014. PMID 24671197
- [Background] Fjeldstad C, Fjeldstad AS, Acree LS, Nickel KJ, Gardner AW. The influence of obesity on falls and quality of life. Dyn Med. 2008 Feb 27;7:4. doi: 10.1186/1476-5918-7-4. PMID 18304350
- [Background] Mitchell RJ, Lord SR, Harvey LA, Close JC. Associations between obesity and overweight and fall risk, health status and quality of life in older people. Aust N Z J Public Health. 2014 Feb;38(1):13-8. doi: 10.1111/1753-6405.12152. PMID 24494939
- [Background] de Souza SA, Faintuch J, Valezi AC, Sant' Anna AF, Gama-Rodrigues JJ, de Batista Fonseca IC, Souza RB, Senhorini RC. Gait cinematic analysis in morbidly obese patients. Obes Surg. 2005 Oct;15(9):1238-42. doi: 10.1381/096089205774512627. PMID 16259878
- [Background] Yeh SH, Chuang H, Lin LW, Hsiao CY, Eng HL. Regular tai chi chuan exercise enhances functional mobility and CD4CD25 regulatory T cells. Br J Sports Med. 2006 Mar;40(3):239-43. doi: 10.1136/bjsm.2005.022095. PMID 16505081
- [Background] Audette JF, Jin YS, Newcomer R, Stein L, Duncan G, Frontera WR. Tai Chi versus brisk walking in elderly women. Age Ageing. 2006 Jul;35(4):388-93. doi: 10.1093/ageing/afl006. Epub 2006 Apr 19. PMID 16624847
- [Background] Yildirim P, Ofluoglu D, Aydogan S, Akyuz G. Tai Chi vs. combined exercise prescription: A comparison of their effects on factors related to falls. J Back Musculoskelet Rehabil. 2016 Aug 10;29(3):493-501. doi: 10.3233/BMR-150645. PMID 26519119
- [Background] Xiang Y, Lu L, Chen X, Wen Z. Does Tai Chi relieve fatigue? A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2017 Apr 5;12(4):e0174872. doi: 10.1371/journal.pone.0174872. eCollection 2017. PMID 28380067
- [Background] Xu F, Letendre J, Bekke J, Beebe N, Mahler L, Lofgren IE, Delmonico MJ. Impact of a program of Tai Chi plus behaviorally based dietary weight loss on physical functioning and coronary heart disease risk factors: a community-based study in obese older women. J Nutr Gerontol Geriatr. 2015;34(1):50-65. doi: 10.1080/21551197.2014.1003672. PMID 25803604
- [Background] Thornton EW, Sykes KS, Tang WK. Health benefits of Tai Chi exercise: improved balance and blood pressure in middle-aged women. Health Promot Int. 2004 Mar;19(1):33-8. doi: 10.1093/heapro/dah105. PMID 14976170
- [Background] Dechamps A, Gatta B, Bourdel-Marchasson I, Tabarin A, Roger P. Pilot study of a 10-week multidisciplinary Tai Chi intervention in sedentary obese women. Clin J Sport Med. 2009 Jan;19(1):49-53. doi: 10.1097/JSM.0b013e318193428f. PMID 19124984
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Topolski TD, LoGerfo J, Patrick DL, Williams B, Walwick J, Patrick MB. The Rapid Assessment of Physical Activity (RAPA) among older adults. Prev Chronic Dis. 2006 Oct;3(4):A118. Epub 2006 Sep 15. PMID 16978493
- [Background] Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S350-70. doi: 10.1002/acr.20538. No abstract available. PMID 22588756
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Lin MR, Hwang HF, Hu MH, Wu HD, Wang YW, Huang FC. Psychometric comparisons of the timed up and go, one-leg stand, functional reach, and Tinetti balance measures in community-dwelling older people. J Am Geriatr Soc. 2004 Aug;52(8):1343-8. doi: 10.1111/j.1532-5415.2004.52366.x. PMID 15271124
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Li F, Harmer P, McAuley E, Fisher KJ, Duncan TE, Duncan SC. Tai Chi, self-efficacy, and physical function in the elderly. Prev Sci. 2001 Dec;2(4):229-39. doi: 10.1023/a:1013614200329. PMID 11833926

RESULTS

PARTICIPANT FLOW:
Groups:
- Tai Chi Intervention: The intervention group received Tai Chi instruction via a weekly group session and home use of a DVD (digital versatile disc) for a period of 8 weeks.
- Control Group: The control group received no formal instruction in physical activity.
Period: Overall Study
Arm/Group | Tai Chi Intervention | Control Group
Started | 11 | 6
Completed | 7 | 5
Not Completed | 4 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Scheduling difficulties | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Tai Chi Intervention: The intervention group received Tai Chi instruction via a weekly group session and home use of a DVD for a period of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Tai Chi Intervention | Control Group | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.6) | 51.8 (10.3) | 51.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Weight [Mean (Standard Deviation); unit: pounds] | 278.36 (28.95) | 266.72 (23.01) | 273.51 (26.18)
BMI [Mean (Standard Deviation); unit: kg/meters squared] | 45.93 (4.9) | 50.04 (3.63) | 47.64 (4.72)
Four Square Step Test [Mean (Standard Deviation); unit: seconds] | 9.91 (2.02) | 10.17 (2.82) | 10.02 (2.27)
30 Second Sit to Stand [Mean (Standard Deviation); unit: repetitions] | 13.14 (2.12) | 13.80 (3.83) | 13.42 (2.81)
Timed Up and Go [Mean (Standard Deviation); unit: seconds] | 8.62 (1.27) | 10.08 (1.67) | 9.23 (1.57)
6 Minute Walk Test [Mean (Standard Deviation); unit: feet] | 416.14 (95.69) | 363.20 (86.76) | 394.08 (92.06)

OUTCOME MEASURES:

1. Primary Outcome: Four Square Step Test
Description: Three-quarter inch diameter plastic tubing was placed on the ground to form a plus sign. The participant was required to step as fast as possible starting in square 1 in a clockwise direction and then returning counterclockwise making full contact in each square with both feet and not touching the tubing. The participants were required to complete the Four Square Step Test in 15 seconds or less in order to be included in the study based on the research that a time longer than 15 seconds is predictive of multiple falls. The results were compared at the conclusion of the study as an indicator of balance.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention 1 | Tai Chi Intervention 2
Number analyzed (Participants) | 7 | 5
seconds
  Pre-test | 9.91 (2.02) | 10.17 (2.82)
  Post-test | 8.93 (2.04) | 9.50 (1.74)

2. Primary Outcome: Zeno Walkway Analysis of Gait Speed
Description: Participants were asked to walk along the gait mat for a total of four passes. A piece of tape was placed one meter before and after the gait mat. Participants were instructed to turn around once they reached the piece of tape to decrease the effects of acceleration and deceleration on the gait mat. Data collected on the Protokinetics Zeno Walkway included the participants' gait speed.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Tai Chi Intervention | Control Group
Number analyzed (Participants) | 7 | 5
meters/second
  Gait Speed Pre Test | 1.20 (.14) | 1.07 (.23)
  Gait Speed Post Test | 1.27 (.14) | 1.17 (.21)

3. Primary Outcome: 36-item Short Form Health Survey (SF-36)
Description: The SF-36 was used to measure how each participant viewed their physical and mental health. The questionnaire contained sections that covered vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Overall, the SF-36 has the ability to measure the well-being of older adults . Scores on the SF-36 range from 0-700, with a lower score identifying greater disability and a higher score suggesting less disability.
Time Frame: 10 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Tai Chi Intervention | Control Group
Number analyzed (Participants) | 7 | 5
score on a scale
  Overall Score, Pre Test | 586.0 [139 to 663] | 564.0 [221.5 to 615]
  Overall Score, Post Test | 598.5 [289 to 680] | 533.0 [247.3 to 644]

4. Primary Outcome: Six Minute Walk Test (6MWT)
Description: The 6MWT is a submaximal test of endurance measuring total distance walked in six minutes. A 100 foot walking path was measured down a level, hard surfaced hallway. The participant was asked to repeatedly walk the complete length of the 100 foot walking path as many times as possible in six minutes at a comfortable pace. The participant was allowed to rest during this test, however, the timer did not stop until the six minute time frame had been completed. The total distance upon completion of the 6MWT was documented.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tai Chi Intervention 1 | Tai Chi Intervention 2
Number analyzed (Participants) | 7 | 5
meters
  Pre-test | 126.84 (29.17) | 110.70 (26.45)
  Post-test | 131.58 (30.81) | 116.52 (25.01)

5. Primary Outcome: 30 Second Sit to Stand
Description: The 30 Second Sit to Stand is a test of lower extremity functional strength. This test consists of rising from a standard height chair and returning to sitting as many times as the person is able to within 30 seconds without the use of their upper extremities. It is a measure of lower extremity functional strength.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Tai Chi Intervention 1 | Tai Chi Intervention 2
Number analyzed (Participants) | 7 | 5
repetitions
  Pre-test | 13.14 (2.12) | 13.80 (3.84)
  Post-test | 13.29 (1.50) | 14.60 (2.70)

6. Primary Outcome: Timed up and go Test
Description: The Timed Up and Go test (TUG) begins with the participant seated in an armchair. The participant is instructed to stand up and walk at a comfortable pace to a mark three meters in front of the chair, turn around, walk back to the chair, and sit down. The test is timed, and participants are allowed to use the arms of the chair and an assistive device if they choose. This assessment correlates with fall risk and functional mobility.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention 1 | Tai Chi Intervention 2
Number analyzed (Participants) | 7 | 5
seconds
  Pre-test | 8.62 (1.27) | 10.08 (1.67)
  Post-test | 8.07 (1.51) | 9.46 (2.91)

7. Primary Outcome: Single Leg Stance Test
Description: The Single Leg Stance test (SLS) test measures static balance while standing on one leg, with a longer time indicating better balance ability. A participant would stand on one leg and hold the position as long as they could up to 30 seconds. Participants were required to perform 3 trials with eyes open and 3 trials with eyes closed on both limbs. The longest of the three trials was used for data analysis. The timer was stopped in the following situations: (1) the foot of the non-stance leg touched the floor, (2) the lower extremities made contact with each other, (3) the participant exceeded 30 seconds of single leg stance, or (4) the participant opened their eyes on the eyes closed trial.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Intervention 1 | Tai Chi Intervention 2
Number analyzed (Participants) | 7 | 5
seconds
  Eyes Closed, Right Pre-test | 1.95 (2.23) | 3.29 (2.23)
  Eyes Closed, Right Post-test | 2.22 (2.32) | 3.62 (1.60)
  Eyes Closed, Left Pre-test | 3.71 (2.29) | 5.27 (4.70)
  Eyes Closed, Left Post-test | 8.35 (10.56) | 3.53 (2.17)

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events during the study period, which was up to 10 weeks for all participants, from the initial data collection point to the final data collection point.
Arm/Group | Tai Chi Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT04106661/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT04106661/ICF_001.pdf